CLINICAL TRIAL: NCT04081519
Title: Stimulation of Parieto-hippocampal Connectivity in Patients With Major Depressive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bonn (Other)
Collaborators: Clemens Mielacher, University Hospital, Bonn (Unknown)
Responsible Party: Principal Investigator, Rene Hurlemann, Chair of the Medical Psychology Division and Deputy Chair of the Department of Psychiatry, University Hospital, Bonn
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SHIP
Record Dates: First submitted 2019-08-27; First posted 2019-09-09 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Depression; Depressive Disorder; Depressive Episode; Depressive Disorder, Major
Keywords: Repetitive Transcranial Magnetic Stimulation; Theta Burst Stimulation; rTMS; TBS; resting-state fMRI; functional connectivity
MeSH Terms: conditions — Depression; Depressive Disorder; Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DLPFC-DLPFC (Active Comparator): 15 sessions of active rTMS over DLPFC + 15 sessions of active rTMS over DLPFC
  Interventions: Device: active rTMS over DLPFC; Device: Add-on active rTMS over DLPFC
- DLPFC-LPC (Experimental): 15 sessions of active rTMS over DLPFC + 15 sessions of active rTMS over LPC
  Interventions: Device: active rTMS over DLPFC; Device: Add-on active rTMS over LPC
- DLPFC-SHAM (Sham Comparator): 15 sessions of active rTMS over DLPFC + 15 sessions of sham rTMS over DLPFC or LPC
  Interventions: Device: active rTMS over DLPFC; Device: Add-on sham rTMS

INTERVENTIONS:
Device: active rTMS over DLPFC — 15 sessions of active rTMS over DLPFC
Device: Add-on active rTMS over DLPFC — 15 additional sessions of active rTMS over DLPFC
  Arms: DLPFC-DLPFC
Device: Add-on active rTMS over LPC — 15 additional sessions of active rTMS over LPC
  Arms: DLPFC-LPC
Device: Add-on sham rTMS — 15 additional sessions of sham rTMS over DLPFC or LPC
  Arms: DLPFC-SHAM

SUMMARY:
This study aims to investigate the effects of individualized repetitive transcranial magnetic stimulation (rTMS) of parieto-hippocampal functional connectivity in patients with major depressive disorder (MDD). Specifically, patients will be randomized to one of three groups and will receive 15 days of rTMS over three weeks. Each day they will receive one active session of rTMS over the dorsolateral parietal cortex (DLPFC) and depending on group assignment another session either A) active rTMS over DLPFC, B) active rTMS over left and right lateral parietal cortex (LPC), or C) sham rTMS over DLPFC or LPC. Stimulation targets in the LPC will be individualized for each patient based on their resting-state functional connectivity between the hippocampus and LPC. Clinical, neuropsychological and fMRI data will be acquired before and after the treatment course.

ELIGIBILITY:
Inclusion Criteria:

* fulfilled criteria for unipolar major depressive disorder for at least four weeks
* did not respond to a minimum of one or did not tolerate a minimum of two antidepressants in the current episode

Exclusion Criteria:

* metal in the brain or the skull
* cardiac pacemaker or intracardiac lines
* medication infusion devices
* heart or brain surgery
* pregnancy
* substance induced depression
* history of substance abuse
* psychotic episodes
* bipolar disorder
* anorexia
* posttraumatic stress disorder (current or within the last 12 months)
* claustrophobia
* any condition resulting in increased intracranial pressure
* traumatic brain injury
* history of epilepsy
* cerebral aneurysms
* dementia
* Morbus Parkinson
* Chorea Huntington
* multiple sclerosis
* stroke or transient ischemic attack (within the last 2 years)
* previous antidepressive treatment with rTMS, electroconvulsive therapy (within the last 3 months), vagus nerve stimulation or deep brain stimulation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2016-08-02 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-06-22 (Actual)

PRIMARY OUTCOMES:
Change in depression severity as measured by the Hamilton Depression Rating Scale (HAMD-17) | Four measurement time points with a seven-day interval starting on the first day of stimulation, and ending three days after the last day of stimulation
  Remission defined as HAMD-17 score (range: 0 to 52, lower scores represent better outcome) of less than or equal to 8 after the rTMS course. Response defined as a reduction of at least 50% from baseline in HAMD-17 score after treatment.
Change in functional connectivity coefficients based on resting-state fMRI | 3 days prior to first rTMS session and 3 days after last rTMS session
  Seed-to-voxel and ROI-to-ROI functional connectivity analysis of rs-fMRI data.
Change in task-based fMRI activation during associative memory paradigm | 3 days prior to first rTMS session and 3 days after last rTMS session
  Functional magnetic resonance imaging (fMRI) will be performed to measure blood-oxygen-level dependent signal encoding and retrieval with a focus on hippocampal regions.

SECONDARY OUTCOMES:
Change in depression severity as measured by the Beck's Depression Inventory (BDI-II) | 3 days prior to first rTMS session and 3 days after last rTMS session, follow-up after 4, 8 and 12 weeks
  Remission defined as BDI-II score (range: 0 to 63, lower scores represent better outcome) of less than or equal to 12 after the rTMS course. Response defined as a reduction of at least 50% from baseline in BDI-II score after treatment.
Change in visual memory as assessed by the Delayed Matching to Sample test (DMS) | 3 days prior to first rTMS session and 3 days after last rTMS session
  Subjects will be assessed in the domain of visual memory by undergoing computorized neurological testing. Outcome varible is percentage of correct answers.
Change in spatial planning as assessed by the One Touch Stockings of Cambridge (OTS) | 3 days prior to first rTMS session and 3 days after last rTMS session
  Subjects will be assessed in the domain of spatial planning by undergoing computorized neurological testing. Outcome varible is the mean number of choices to correct answer.
Change in visual sustained attention as assessed by the Rapid Visual Information Processing (RVP) | 3 days prior to first rTMS session and 3 days after last rTMS session
  Subjects will be assessed in the domain of visual sustained attention by undergoing computorized neurological testing. Outcome varible is the target sensitivity A'.
Change in working memory as assessed by the Spatial Working Memory (SWM) | 3 days prior to first rTMS session and 3 days after last rTMS session
  Subjects will be assessed in the domain of working memory by undergoing computorized neurological testing. Outcome varible is the total number of errors.
Change in task-based fMRI activation during social touch paradigm | 3 days prior to first rTMS session and 3 days after last rTMS session
  Functional magnetic resonance imaging (fMRI) will be performed to measure blood-oxygen-level dependent signal while participants receive tactile stimulation.
Change in task-based fMRI activation during emotional processing paradigm | 3 days prior to first rTMS session and 3 days after last rTMS session
  Functional magnetic resonance imaging (fMRI) will be performed to measure blood-oxygen-level dependent signal while participants perform an emotional processing task.

CONTACTS AND LOCATIONS:
Overall Officials: René Hurlemann, Prof., Principal Investigator — University Hospital, Bonn
Locations (1):
- Klinik und Poliklinik für Psychiatrie und Psychotherapie, Bonn, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fox MD, Buckner RL, White MP, Greicius MD, Pascual-Leone A. Efficacy of transcranial magnetic stimulation targets for depression is related to intrinsic functional connectivity with the subgenual cingulate. Biol Psychiatry. 2012 Oct 1;72(7):595-603. doi: 10.1016/j.biopsych.2012.04.028. Epub 2012 Jun 1. PMID 22658708
- [Background] Wang JX, Rogers LM, Gross EZ, Ryals AJ, Dokucu ME, Brandstatt KL, Hermiller MS, Voss JL. Targeted enhancement of cortical-hippocampal brain networks and associative memory. Science. 2014 Aug 29;345(6200):1054-7. doi: 10.1126/science.1252900. PMID 25170153
- [Background] Blumberger DM, Vila-Rodriguez F, Thorpe KE, Feffer K, Noda Y, Giacobbe P, Knyahnytska Y, Kennedy SH, Lam RW, Daskalakis ZJ, Downar J. Effectiveness of theta burst versus high-frequency repetitive transcranial magnetic stimulation in patients with depression (THREE-D): a randomised non-inferiority trial. Lancet. 2018 Apr 28;391(10131):1683-1692. doi: 10.1016/S0140-6736(18)30295-2. Epub 2018 Apr 26. PMID 29726344
- [Background] Lefaucheur JP, Andre-Obadia N, Antal A, Ayache SS, Baeken C, Benninger DH, Cantello RM, Cincotta M, de Carvalho M, De Ridder D, Devanne H, Di Lazzaro V, Filipovic SR, Hummel FC, Jaaskelainen SK, Kimiskidis VK, Koch G, Langguth B, Nyffeler T, Oliviero A, Padberg F, Poulet E, Rossi S, Rossini PM, Rothwell JC, Schonfeldt-Lecuona C, Siebner HR, Slotema CW, Stagg CJ, Valls-Sole J, Ziemann U, Paulus W, Garcia-Larrea L. Evidence-based guidelines on the therapeutic use of repetitive transcranial magnetic stimulation (rTMS). Clin Neurophysiol. 2014 Nov;125(11):2150-2206. doi: 10.1016/j.clinph.2014.05.021. Epub 2014 Jun 5. PMID 25034472
- [Background] Daumann J, Fischermann T, Heekeren K, Henke K, Thron A, Gouzoulis-Mayfrank E. Memory-related hippocampal dysfunction in poly-drug ecstasy (3,4-methylenedioxymethamphetamine) users. Psychopharmacology (Berl). 2005 Aug;180(4):607-11. doi: 10.1007/s00213-004-2002-8. Epub 2005 Sep 14. PMID 15372137